CLINICAL TRIAL: NCT07138170
Title: Comparison of Distal and Proximal Radial Artery Patency Following Coronary Catheterization, A Real Look at a Special Community: An Open Randomized Clinical Trial
Brief Title: Comparison of Distal and Proximal Radial Artery Patency Following Coronary Catheterization, A Real Look at a Special Community
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordanian Research and Artificial Intelligence Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RAPT
Record Dates: First submitted 2025-08-10; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Radial Artery Occlusion Following Coronary Catheterization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The ultrasound operator is blinded to the group of the patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal Radial Artery Access Group (Experimental)
  Interventions: Procedure: Proximal Radial Artery Access
- Distal Radial Artery Access Group (Experimental)
  Interventions: Procedure: Distal Radial Artery Access

INTERVENTIONS:
Procedure: Proximal Radial Artery Access — Using Proximal Radial Artery Access for Cardiac Catheterization
  Arms: Proximal Radial Artery Access Group
Procedure: Distal Radial Artery Access — Using Distal Radial Artery access for Cardiac Catheterization
  Arms: Distal Radial Artery Access Group

SUMMARY:
Background: Radial artery occlusion is the Achilles' heel of radial artery catheterization; this well-known complication is very serious, with an incidence ranging between 5-30% when using the proximal or anterior radial artery access. Emerging evidence suggests that distal radial access may preserve radial artery patency more effectively, with reported occlusion rates between one and two percent. Maintaining radial artery patency is crucial for future procedures, such as utilizing the radial artery as a conduit for CABG (Coronary Artery Bypass Grafting) or for shunts in dialysis patients.

Objective: The aim of this study is to compare distal and proximal radial artery access in patients undergoing coronary catheterization by evaluating radial artery patency and complication rates at time zero(1-2 days post-procedure), and at 1-6 months post-procedure. This is the first randomized clinical trial of its kind conducted in Palestine and possibly the broader Middle East region, where resources are often very limited, which in turn will reflect a real look at some real communities' experiences.

Methods: This randomized clinical trial will include 250 patients over eighteen years old who are scheduled for coronary catheterization. Participants will be randomly assigned either to proximal radial artery access or distal radial artery access. This approach created two equal groups: one group undergoing distal radial artery access and the other proximal radial artery access, with one hundred twenty-five patients in each group. Due to the nature of our practice in the two cardiac centers sharing in the study, all procedures will be performed by very experienced interventional cardiologists. Radial artery patency will be evaluated by a blinded ultrasound specialist at 1-2 days and at 1-6 months post-index procedure. Complication rates, including pain, bleeding, hematoma, and hand function, will also be assessed as secondary outcomes. In cases where radial access is unsuccessful, crossover to an alternative access site, such as the contralateral radial or femoral artery, will be documented.

Expected Results: It is hypothesized that distal radial access will result in significantly lower rates of radial artery occlusion compared to proximal access across the two time points. Complication rates are also expected to be lower in the distal radial artery group..

Conclusion: This study may support the use of distal radial access as a preferred approach in coronary catheterization due to improved long-term radial artery patency, without an increase in access-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults above the age of 18 years old and accepting participation in the study.

Exclusion Criteria:

* patients below the age of 18 or declined to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Radial Artery occlusion | 1-2 days and 1-6 months post procedure

SECONDARY OUTCOMES:
Number of participants with Pain | 1-2 days and 1-6 months post-procedure.
  The patients will be asked to rate their pain on a 1-10 scale.
Number of patients with bleeding | 1-2 days and 1-6 months post-procedure.
  the presence of bleeding will be assed by physical examination of the access site
Number of Participants with hematoma | 1-2 days and 1-6 months post-procedure.
  The presence of hematoma will be assessed by physical examination of the access site
sensory and motor hand function | 1-2 days and 1-6 months post-procedure.
  Sensory and motor hand function will be assessed by physical examination of the hand
Number of patients with unsuccessful radial access | At the time of procedure
  In cases where radial access is unsuccessful, crossover to an alternative access site, such as the contralateral radial or femoral artery, will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Izraiq, Medical Doctor, Principal Investigator — The Specialty Hospital; Raed Aqel, Medical Doctor, Principal Investigator — Al-Mezan Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinha SK, Jha MJ, Mishra V, Thakur R, Goel A, Kumar A, Singh AK, Sachan M, Varma CM, Krishna V. Radial Artery Occlusion - Incidence, Predictors and Long-term outcome after TRAnsradial Catheterization: clinico-Doppler ultrasound-based study (RAIL-TRAC study). Acta Cardiol. 2017 Jun;72(3):318-327. doi: 10.1080/00015385.2017.1305158. Epub 2017 Mar 30. PMID 28636520